CLINICAL TRIAL: NCT06567795
Title: Prospective, Multi-center, Longitudinal, Study for PRimary IndividualiZed Evaluation of Cardiovascular Events in Patients With Diabetes Mellitus Using hemoTAG
Brief Title: PRimary IndividualiZed Evaluation of Cardiovascular Events in Patients With Diabetes Mellitus Using hemoTAG
Acronym: PRIZETAG
Status: Recruiting | Type: Observational
Sponsor: Aventusoft, LLC. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HT-101-VV-032; R44HL149561-03 (NIH)
Record Dates: First submitted 2024-05-21; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus Type 2; Cardiovascular Diseases; Coronary Artery Disease; Cerebrovascular Disease; Peripheral Artery Disease
Keywords: Diabetes Mellitus; Cardiovascular Diseases; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Coronary Artery Disease; Cerebrovascular Disorders; Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- HEMOTAG with Standard of Care in DM patients: HEMOTAG with Standard of Care: To evaluate the proportion of diabetic mellitus patients with cardiovascular events as identified by HEMOTAG measurements over a 12 month duration.
  Interventions: Device: Hemotag

INTERVENTIONS:
Device: Hemotag — Hemotag non-invasive medical device is used to see cardiac function for DM2 patients at-home for 30 days

SUMMARY:
To evaluate the proportion of diabetic mellitus patients with CV events as measured by HEMOTAG.

DETAILED DESCRIPTION:
This is a prospective, multi-center, longitudinal study to evaluate the proportion of cardiovascular events in diabetic mellitus patients identified by HEMOTAG evaluations, utilizing cardiac time interval measurements being treated in outpatient clinics. An enriched diabetic patient population, currently undergoing standard medical care for their diabetes management (per the American Diabetes Association) will be invited to participate within this study. All patients will complete their standard of care assessments including, vital signs, creatinine, eGFR, fasting Cholesterol (including HDL and LDL), HbA1c,and NT-pro BNP, at their regularly scheduled diabetic clinic visits. During the enrollment visit, patients will undergo a baseline HEMOTAG evaluation, cardiovascular event assessment as well as baseline questionnaire assessments. Patients will be shipped a HEMOTAG device with electrodes, and HEMOTAG measurements will be conducted at least three days a week for a 30-day period at-home. This will occur after the Baseline Visit, after the 6-month Visit, and following any hospitalizations due to cardiac events during the 12-month study.

All patients will undergo standard of care follow-up visits at their normal 6 month and 12 month visits and will repeat the HEMOTAG evaluation (in clinic), cardiovascular event assessment, NT-pro BNP, as well as questionnaire assessments. Results of standard of care assessments including, vital signs, creatinine, eGFR, fasting Cholesterol (including HDL/LDL),and HbA1c, will be collected if performed during their regularly scheduled diabetic clinic visits. Throughout the course of this study, all study participant's medical records will reviewed and assessed for the occurrence of cardiac events (including hospitalizations, emergency room visits/urgent care visits, other cardiac assessments, and death) for up to 12 months. Results from cardiac testing (examples: Echo, Cardiac Catheterization, Stress Tests, etc) that may occur during the 12-month monitoring period will be collected as part of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients older than 40 years of age.
2. Diagnosis of Type 2 Diabetes Mellitus (insulin dependent or non-insulin dependent) for at least 5 years.
3. Diagnosis of Cardiovascular Disease (Coronary Artery Disease, Cerebrovascular Disease, Peripheral Artery Disease, etc…) --OR--

   Have one (1) of the following concomitant medical diagnoses:
   1. Diabetic Retinopathy (proliferative or non-proliferative)
   2. Diabetic Nephropathy (eGFR <60 mL/min/1.73m2 and/or urine albumin/creatinine ratio ≥30 mg/g)
   3. Diabetic Neuropathy
   4. Elevated High-sensitivity C-reactive protein (hs-CRP) --AND--

      Have a history of two (2) or more of the following:
   5. Diagnosis of Hypertension for at least 6 months or more (treated or untreated)
   6. Hypercholesterolemia (LDL-C >100 mg/dL)
   7. Obesity (Body Mass Index (BMI) ≥ 27 for men or ≥ 22 for women)
   8. History of Smoking
4. Willingness to undergo HEMOTAG evaluation.
5. Willingness to undergo Standard of Care visits/assessments and NT-pro BNP lab evaluations.
6. Willingness to conduct at-home HEMOTAG evaluations at least three days per week within a 30-day time period after the completion of the Baseline Visit, after the 6 month visit and following discharge from any hospitalizations due to a cardiac events during the 12 month study period.
7. Willingness to receive and return shipping of the HEMOTAG KIT at each time point as required by the protocol
8. Able to give informed consent.

Exclusion Criteria:

1. Terminal condition with life expectancy less than 12 months as determined by investigator.
2. Physical deformity in the chest area or lesion that may prevent proper HEMOTAG application or adjustment.
3. Illness/ Condition which may be aggravated or cause significant discomfort to the patient by the application of the HEMOTAG (skin issues, e.g. Intolerance to use of skin electrodes).
4. Participant enrolled in another interventional study (observational or registries are not excluded).
5. Prisoners and wards of the state.
6. Impaired cognitive ability or any other state that may prevent full compliance with the study protocol, according to investigator's assessment.
7. Participants unable to provide informed, voluntary decision to participate in research study as determined by the investigator. (Exclude participants who necessitate the involvement of a legally authorized representative.)
8. Inability to provide informed consent (Must speak English).
9. Women who are pregnant or are planning to become pregnant during the study.
10. Women of childbearing potential who are unwilling or unable to comply with contraception measures.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients that meet inclusion exclusion criteria
Sampling Method: Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2027-03-18 (Estimated)

PRIMARY OUTCOMES:
To evaluate the proportion of diabetic mellitus patients with cardiovascular events as identified by HEMOTAG measurements over a 12 month duration. | 12 months
  The primary endpoint will be to evaluate CV events measured by a composite endpoint defined by unplanned hospitalizations, emergency room visits/urgent care visits (that do not result in hospitalization), for cardiovascular events or death within the observation period of 12 months.

SECONDARY OUTCOMES:
Secondary objective will evaluate various cardiac events occurring over time throughout the observational period as well as quality of life measurements for 6 months. | 6 months
  Composite endpoint consisting of unplanned hospitalizations, emergency room visits/urgent care visits (that do not result in hospitalization), for cardiovascular events or death within the observation period of 6 months.
Correlation of AO and CE at 6 and 12 months | 12 months
  Correlation of AO and CE at 6 and 12 months
Correlation of CTI and CE at 6 and 12 months | 12 months
  Correlation of CTI and CE at 6 and 12 months
All Deaths for 12 months | 12 months
  All Deaths for 12 months
Median time to composite of worsening left ventricular dysfunction or heart failure among diabetic patients at 6 months and 12 months | 12 months
  Median time to composite of worsening left ventricular dysfunction or heart failure among diabetic patients at 6 months and 12 months
Six Minute Walk Test (Borg Dyspnea/Borg Fatigue Scale) | 12 months
  Six Minute Walk Test (Borg Dyspnea/Borg Fatigue Scale) Excellent: Distance is typically above 700 meters. Good: Distances within the average range between 400 and 700 meters Poor: Distances below the average range, indicating potential limitations in aerobic capacity and functional status is below 400 meters.
Median time to heart failure at 6 and 12 months | 12 months
  Median time to heart failure at 6 and 12 months
Median time to Left Ventricular Dysfunction at 6 and 12 months | 12 months
  Median time to Left Ventricular Dysfunction at 6 and 12 months
Health State as measured by the EQ5D5L ( EuroQol 5 Dimensions 5 Levels) | 12 months
  Health State as measured by the EQ5D5L: 1 is the best possible value (indicating no problems), and 5 is the worst (indicating extreme problems).
  1. indicates no problems
  2. indicates slight problems
  3. indicates moderate problems
  4. indicates severe problems
  5. indicates extreme problems

OTHER OUTCOMES:
All cause hospitalizations | 12 months
  All cause hospitalizations
Health Status as measured by the LVD-36 | 12 months
  Health Status as measured by the LVD-36 Low Scores: Indicate fewer symptoms and better quality of life. High Scores: Indicate more severe symptoms and poorer quality of life.
Productivity questionnaire | 12 months
  Productivity questions deal with how health issues or their treatment have affected the subject's ability to remain in the workforce and perform daily activities in the home.
Health care resource utilization | 12 months
  Health care resource utilization Frequency of visits to the emergency department within 30 days Rates of patients being readmitted to the hospital within a 30 day time period. Reporting of outpatient visits within 30 days
Treatment Satisfaction | 12 months
  Treatment Satisfaction: Responses are rated on a 7-point scale, ranging from 1 (extremely dissatisfied) to 7 (extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Metabolic Research Institute, Inc, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: website — https://aventusoft.com